CLINICAL TRIAL: NCT01984099
Title: The Efficacy of Methotrexate for the Prevention of Postmolar Gestational Trophoblastic Disease Among Patients With High-Risk Hydatidiform Mole
Brief Title: RCT on the Efficacy of Methotrexate for the Prevention of GTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH 2009-044
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Hydatidiform Mole
Keywords: Postmolar Gestational Trophoblastic Disease, Hydatidiform Mole
MeSH Terms: conditions — Hydatidiform Mole | interventions — Methotrexate; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoprohylaxis Group (Active Comparator): Chemoprohylaxis Group: the treatment group, will be given a single course of methotrexate within fourteen days from molar evacuation. Methotrexate will be given at 0.4 mg/kg intramuscularly per day for 5 days. No chemotherapy will be administered if the hemoglobin is lower than 10 g/L, WBC is less than 3.0 x 10 g/L or more than 10.0 x 10 g/L, absolute neutrophil count is less than 1.5, platelet count is lower than 100,000/cu.cc., patient has elevated liver and renal function test and has concurrent infection.
  Interventions: Drug: Methotrexate
- Control Group (Placebo Comparator): Control Group: will be given a placebo in a form of Vitamin B Complex (Bee ALL), intramuscularly or intravenously.
  Interventions: Drug: Vitamin B Complex

INTERVENTIONS:
Drug: Methotrexate — Patients will be given a single course of methotrexate within fourteen days from molar evacuation.
  Arms: Chemoprohylaxis Group
Drug: Vitamin B Complex — Patients will be given a placebo in a form of Vitamin B Complex (Bee ALL), intramuscularly or intravenously.
  Other Names: Bee ALL
  Arms: Control Group

SUMMARY:
A randomized, controlled trial to evaluate the efficacy of methotrexate for the prevention of postmolar gestational trophoblastic disease among patients with high-risk hydatidiform mole.

DETAILED DESCRIPTION:
A randomized, controlled trial to evaluate the efficacy of methotrexate for the prevention of postmolar gestational trophoblastic disease among patients with high-risk hydatidiform mole.

Women who will undergo suction curettage for complete hydatidiform mole at the Philippine General Hospital, who are at risk for developing postmolar gestational trophoblastic disease will be included in the study. Patients will receive either a single course of methotrexate or vitamin B complex (Benutrex) within fourteen days from molar evacuation. Patients' serum beta HCG will be monitored 1 week after molar evacuation and then every 2 weeks until the titers become normal for three consecutive determinations, then monthly for 6 months (every 2 months for the next 6 months).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis and molar evacuation done at the Department of Obstetrics and Gynecology of the Philippine General Hospital;
* patients who will undergo suction curettage for evacuation of molar pregnancy;
* histopathologically confirmed complete hydatidiform mole;
* must have at least one of the following risk factors for the development of postmolar gestational trophoblastic disease:

  * uterine size larger than age of gestation of more than 6 weeks
  * serum B-hCG titer more than or equal to 100,000 mlU/ml
  * theca lutein cysts more than or equal to 6 cms in size
  * gravidity of 4 or more
  * recurrent molar pregnancy
  * medical complications arising from trophoblastic proliferation such as DIC, pre-eclampsia, thyrotoxicosis, pulmonary insufficiency
* complete data;
* patient must have at least one year of regular follow-up and hCG monitoring following onset of remission;
* should have signed the consent form.

Exclusion Criteria:

* patients who are lost to follow-up or with incomplete data
* patients who underwent total hysterectomy for evacuation of molar pregnancy
* patients who are unable to complete the methotrexate treatment
* patients who get pregnant within a year following remission
* patients with a previous history of gestational trophoblastic neoplasia
* patients with medical problems/complications that inhibit administration of methotrexate

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Elevated HCG Level | 4-14 weeks
  1. Diagnosis of postmolar gestational trophoblastic diseases will be based on the occurrence of any of the following conditions:
     * high level of hCG more than 4 weeks post-evacuation (serum level of 20,000mlU/m)
     * progressively increasing or plateuing hCG values at any time after evacuation (minimum of 3 weekly determinations)
     * clinical or histologic evidence of metastasis at any site
     * persistently elevated hCG titer at 14 weeks post-evacuation
     * elevation of previously normal hCG titer after evacuation provided the diagnosis of pregnancy is excluded
  2. Toxicity brought about by the administration of methotrexate will be graded based on the WHO toxicity scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes L. Soriano-Estrella, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- Philippine General Hospital, University of the Philippines Manila, Taft Avenue, Ermita, Manila, Manila, Philippines